CLINICAL TRIAL: NCT01822743
Title: A Single Blind Cross Over Trial to Compare Osteopathic Compression of Pterygopalatine Node to Sham in Patients With Obstructive Sleep Apnea Syndrome and in Healthy Subjects
Brief Title: Osteopathy and Obstructive Sleep Apnea Syndrome II
Acronym: OSTEOSAOSII
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: P111007
Record Dates: First submitted 2013-03-28; First posted 2013-04-02 (Estimated); Last update posted 2022-01-25 (Actual); Status verified 2014-06

CONDITIONS: Obstructive Sleep Apnea Syndrome
Keywords: Osteopathy; Sleep Apnea Syndromes; Obstructive Sleep Apnea; Pcrit; Polysomnography
MeSH Terms: conditions — Sleep Apnea, Obstructive; Sleep Apnea Syndromes | interventions — Manipulation, Osteopathic

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Osteopathic manipulative treatment (Experimental): Osteopathic compression of pterygopalatine node
  Interventions: Procedure: Osteopathic manipulative treatment
- Sham comparator (Sham Comparator): sham Osteopathic pterygopalatine node compression
  Interventions: Procedure: sham comparator

INTERVENTIONS:
Procedure: Osteopathic manipulative treatment — Osteopathic compression of pterygopalatine node
  Arms: Osteopathic manipulative treatment
Procedure: sham comparator
  Arms: Sham comparator

SUMMARY:
The main objective is to evaluate an osteopathic compression of pterygopalatine node in healthy subjects and patients suffering from obstructive apnea syndrome (OSA).

DETAILED DESCRIPTION:
Osteopathic compression will be compared to a sham manoeuvre in a cross over design on apnea hypopnea index, pharyngeal collapsibility and symptoms in patients suffering from OSA, and on symptoms and pharyngeal collapsibility in healthy subjects.

ELIGIBILITY:
Obstructive sleep apnea syndrome patient:

Inclusion criteria :

* Male or Female aged 18 years or more
* Obstructive sleep apnea syndrome with apnea/hypopnea index > or = 15/hour
* Body mass Index <40kg/m2

Exclusion criteria :

* Pregnant or lactating women
* Participating to another trial
* Acute infectious disease of upper respiratory airway tract at inclusion
* Complete nasal obstruction
* Facial neuralgia at inclusion
* Patients not able to stop treatment for OSA within one week before each visit
* Allergy to latex
* Dental extraction within 15 days before inclusion
* Pharyngeal surgery in the past
* Incapable adult
* Patients treated with Selective Serotonin Reuptake Inhibitor

Healthy Volunteers

Inclusion criteria :

* Male or Female aged ≥18 and ≤ 40 years
* No obstructive sleep apnea syndrome
* Body mass Index <30kg/m2
* No chronicle respiratory, neurological, cardiac or able to deteriorate sleep quality disease
* Low obstructive sleep apnea syndrome probability measured with Berlin Scale

Exclusion criteria :

* Pregnant or lactating women
* Participating to another trial
* Acute infectious disease of upper respiratory airway tract at inclusion
* Complete nasal obstruction
* Facial neuralgia at inclusion
* allergy to latex
* dental extraction within 15 days before inclusion
* pharyngeal surgery in the past
* incapable adult
* patients treated background treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2012-01; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Apnea-hypopnea index | 24 hours

SECONDARY OUTCOMES:
Pharyngeal sensitivity test | 30 min
Determination of pharyngeal critical pressure | 24 hours
Daily clinical symptoms of osa | 7 days
Pharyngeal sensitivity test | 24 hours
Determination of pharyngeal critical pressure | 30 min
Inspiratory nasal pic flow | 30 min
Inspiratory nasal pic flow | 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Valérie Attali, MD, Principal Investigator — APHP
Locations (1):
- Service des pathologies du sommeil, Pitié-Salpêtrière hospital, Paris, France

REFERENCES:
- [Result] https://www.mdpi.com/1421774